CLINICAL TRIAL: NCT06358027
Title: Evaluation of the Effects of Different Ventilation Modes Used During Anesthesia Awakening on the Frequency of Postoperative Atelectasis by Lung Ultrasonography: A Prospective Observational Study
Brief Title: Evaluation of the Effects of Different Ventilation Modes Used During Anesthesia Awakening on the Frequency of Postoperative Atelectasis
Status: Not yet recruiting | Type: Observational
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Busra Otlu, Assistant professor, Dokuz Eylul University
Other Study IDs: DokuzEU-ACC-BOtlu-01
Record Dates: First submitted 2024-04-05; First posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Atelectasis, Postoperative Pulmonary
Keywords: Lung Ultrasonography; Atelectasis; Postoperative Pulmonary Complications; Pressure Support Ventilation
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- pressure support ventilation group: when the patients were ready for extubation, anesthesia was terminated by one of the selected pressure support ventilation
  Interventions: Diagnostic Test: lung ultrasound
- manual ventilation group: when the patients were ready for extubation, anesthesia was terminated by one of the selected manual ventilation wake-up methods at the initiative of the relevant anesthesiologist.
  Interventions: Diagnostic Test: lung ultrasound

INTERVENTIONS:
Diagnostic Test: lung ultrasound — The patients included in the study underwent lung imaging with lung ultrasound score twice, in the preoperative preparation room and in the postoperative recovery unit.Both lungs were determined as anterior and posterior axillary lines as anatomical markers and divided into a total of 12 regions, 4 in the anterior thoracic wall, 4 in the lateral wall, and 4 in the posterior region. In our study, we will use the modified LUS scoring, which has been shown to be more sensitive in the diagnosis of postoperative atelectasis in the recovery unit, based on existing literature reviews. The degree of the atelectasis will be determined according to do modified lung ultrasound score. Lung ultrasound score imaging of all patients was performed by the same anesthesiologist.
  Other Names: Modified Transthoracic Ultrasound Scoring System

SUMMARY:
In our study, we aimed to detect atelectasis developing in patients undergoing surgery under general anesthesia using transthoracic lung ultrasonography and to investigate the effect of ventilation methods used during recovery from anesthesia on the formation of postoperative atelectasis.

DETAILED DESCRIPTION:
Postoperative atelectasis is one of the most common pulmonary complications seen in surgical patients. Postoperative pulmonary complications and possible respiratory side effects have long been associated with anesthesia. Pulmonary complications are an important cause of morbidity and mortality in the postoperative period. The incidence of postoperative pulmonary complications due to long-term anesthesia varies between 5% and 80%, depending on the patient population, the surgery performed, and the criteria used to define the complication. It is known that the recovery period makes a significant contribution to the total amount of postoperative atelectasis. Spontaneously breathing patients are under the influence of anesthetic agents and neuromuscular blockers and cannot regain their functional residual capacity. For this reason, it is emphasized that atelectasis may develop in the postoperative period in cases whose anesthesia application is terminated by applying a spontaneous breathing period. Pressure support ventilation (PSV) is widely used for ventilator weaning in the intensive care unit (ICU) and has recently been available on anesthesia machines.

It is expected that the use of lung ultrasonography in operating rooms can reduce the complications that may develop in the postoperative period with evidence-based detection and early postoperative detection of atelectasis in the early postoperative period.

In this study, it was aimed to compare the effect of pre-extubation ventilation mode applied by anesthesia practitioners with ultrasound in the postoperative period on the frequency of atelectasis in adult patients who underwent surgery and whose lungs were evaluated as normal by ultrasound in the preoperative observation room. Modified LUS scores were used as lung ultrasonography evaluation criteria in the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing general anesthesia with supine position
* Endotracheal intubations and mechanical ventilation during general anesthesia
* Operation time is more than 2 hours

Exclusion Criteria:

* Patients who will undergo surgical intervention under emergency conditions
* Pregnancy
* Upper respiratory tract disease in the last 3 weeks
* Previous lung surgery
* Advanced cardiac and/or pleural lung disease and chest wall deformity, and primary or metastatic lung cancer

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patients 18 years of age or older and American Society of Anesthesiologists (ASA) physical status I and III who were scheduled for general anesthesia were included in this prospective observational study.
Sampling Method: Non-Probability Sample
Enrollment: 278 (Estimated)
Dates: Start 2024-04-05 (Estimated); Primary Completion 2024-04-21 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Modified Transthoracic Ultrasound Score | two weeks
  Both lungs were determined as anterior and posterior axillary lines as anatomical markers and divided into a total of 12 regions, 4 in the anterior thoracic wall, 4 in the lateral wall, and 4 in the posterior region. While the anterior and lateral regions were examined in the supine position by placing the probe perpendicular to the thoracic wall and longitudinal in the intercostal spaces with the bat sign displayed, especially the posterior regions close to the diaphragm were examined by placing the probe transversely in the intercostal spaces by turning the patient opposite. According to the systematic LUS protocol, each patient was evaluated for approximately 10-15 minutes and optimum images were obtained.Each area was scored on a scale of 0-3 according to the degree of atelectasis, and a total score between 0 (normal lung ventilation image) and 36 (total loss of ventilation) was calculated.

IPD SHARING:
Plan to Share IPD: No